CLINICAL TRIAL: NCT06325384
Title: VISION-Real World Evaluation
Brief Title: Real World Evaluation of Lifelight®: A Contactless Vital Signs Monitor for Self-monitoring Blood Pressure and Its Comparison to Standard of Care
Acronym: VISION-RWE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xim Limited (Industry)
Collaborators: Barts & The London NHS Trust (Other); Mind Over Matter Medtech Ltd (Industry); Health Innovation Wessex (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRAS ID:321955
Record Dates: First submitted 2024-01-24; First posted 2024-03-22 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cuff Arm (Active Comparator): Blood Pressure Cuff
  Interventions: Device: Blood Pressure Cuff
- LifeLight Arm (Experimental): Contactless Vital Signs Monitor using RPPG
  Interventions: Device: Lifelight

INTERVENTIONS:
Device: Lifelight — Contactless Vital Signs Measurement via RPPG
  Arms: LifeLight Arm
Device: Blood Pressure Cuff — Standard Blood Pressure Cuff Digital
  Arms: Cuff Arm

SUMMARY:
A randomised controlled trial for comparison of real-world feasibility and clinical outcomes of two different methods of home blood pressure monitoring Participants aged 18 years or over with diagnosed and treated hypertension (including via lifestyle interventions) that is not controlled (i.e. in-clinic measurement is 140/90 mmHg or greater) will be recruited from hypertension hospital clinics

DETAILED DESCRIPTION:
Suitable patients from the BHT hypertension clinic patient database will be invited to take part in the study, resulting in the recruitment of 500 people aged 18 years or over who have a clinical diagnosis of hypertension that is treated (including via lifestyle interventions) but not controlled (≥140/90mmHg in-clinic measurement of BP). Study nurses at BHT will facilitate this recruitment and randomise participants to either Lifelight® or BP cuff arm using a secure web-based system in 1:1 ratio, minimised on baseline BP, gender, and BP target (standard hypertension, older hypertension and diabetes). They will also collect all baseline study data, including baseline BP measurements.

The HBPM schedule that all participants will be asked to follow for the full 6-month study duration is HBPM using BP cuff or Lifelight® (depending on into which arm of the study they have been randomised) twice in a sitting for two sittings a day for one week every month. All participants will be asked to record their adherence to HBPM in the provided diary (recording the number of repeat measurements made on each day that those measurements are made and notes about any measurement failures). They will also be requested to record in their diary information about their healthcare resource use (GP appointments, outpatients' appointments, hospitalisations, medication and dose changes, medication adherence) and feedback about their HBPM method every month. All participants will also be asked to complete a set of tailored and validated questionnaires in the provided questionnaire booklet: quality of life.

The diaries and questionnaire booklets include instructions to assist with their accurate completion by participants. Participants will be issued with two diaries during their study participation: one at the baseline visit and one at the 3-month visit. They should complete the diary every day that they are doing HBPM. Participants will be issued with 3 questionnaire booklets during their study participation: two at the baseline visit and one at the 3-month visit. They should complete one questionnaire booklet within one week of their baseline visit, the second booklet within one week of their 3-month visit, and the third booklet within one week of their 6-month visit. Participants will be requested to bring back the diary and questionnaire booklet(s) at their subsequent study visit at BHT. Participants randomised to the Lifelight® arm will be prompted via the app to monitor their BP during the relevant weeks.

People eligible to take part in this study will be adults (18+ years old) with treated but uncontrolled hypertension. People with uncontrolled hypertension have the highest risk of CVD events and therefore the value of HBPM could be greatest for these people. The TASMIN and HOME BP studies focussed on this sub-population of patients with hypertension too, suggesting that future guidelines may continue to provide no recommendation of frequent HBPM for people with controlled hypertension, but a change to the guidelines for people with uncontrolled hypertension.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Established diagnosis of hypertension
* Uncontrolled hypertension defined as office blood pressure ≥140/90mmHg.
* Patients who are pharmacologically treated for their hypertension should have been on stable medication for at least 4 weeks.
* Ability to read, write and understand English to complete the study.
* Capacity to give free, valid informed consent.
* A compatible device that supports Lifelight®, as per xim Ltd.'s constantly updating list of compatible devices. If this is not possible, xim Ltd, might provide a similar device for the purpose of the study.

Exclusion Criteria:

* Patients with stage III hypertension with office blood pressure ≥180/120mmHg or it is unsafe to keep them in the study, in the opinion of the investigators.
* Individuals with diagnosed atrial fibrillation.
* Patients with significant arrhythmias such as SVT (Supraventricular tachycardia) or any rhythm that has significant impact on their BP, poor perfusion, pregnancy, pre-eclampsia, deformities or abnormalities which may prevent proper application of a BP cuff, or skin disorders (anaemia, jaundice, rosacea, psoriasis, acute acne, and erythropoietic protoporphyria)
* Participants who are unwilling to undertake self-monitoring or lacking capacity.
* Partners or spouses of individuals already randomised in the trial
* Patients on dialysis or known ESRD (End-stage kidney disease)
* Patients on active cancer treatment
* Terminally ill patients
* Patients who cannot tolerate sitting for up to one hour.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure Measurement Non Inferiority | 3 Months
  Demonstrate non-inferiority of Lifelight® HBPM compared to cuff-based HBPM for achieving blood pressure control. (5 mmHg non-inferiority margin)

SECONDARY OUTCOMES:
Adherance to Blood Pressure Measurement | 6 Months
  Determine acceptability and adherence of Lifelight® for HBPM in comparison to cuff-based HBPM methods.

CONTACTS AND LOCATIONS:
Locations (1):
- William Harvey Heart Centre, Queen Mary Queen Mary University of London, Charterhouse Square,, London, United Kingdom